CLINICAL TRIAL: NCT05429489
Title: Comparison of the Efficacy of Bilevel Erector Spinae Plane Block and Single Level Erector Spinae Plane Block Versus General Anesthesia in Breast Cancer Surgeries
Brief Title: Erector Spinae Plane Block Versus General Anesthesia in Breast Cancer Surgeries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Institute, Egypt (Other)
Responsible Party: Principal Investigator, Walaa Youssef Elsabeeny, Assistant professor of Anesthesia and Pain management, National Cancer Institute, Egypt
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AP2205-5015
Record Dates: First submitted 2022-06-17; First posted 2022-06-23 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Analgesia
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Bilevel erector spinae plane block (Experimental): Bilevel erector spinae block at 3rd and 5th thoracic vertebral levels
  Interventions: Procedure: Bilevel erector spinae plane block
- Single level erector spinae plane block (Experimental): single level erector spinae plane block at 5th thoracic vertebral levels
  Interventions: Procedure: Single level erector spinae plane block
- Intravenous morphine (Active Comparator): Intravenous morphine 0.1 mg/ kg
  Interventions: Drug: Intravenous morphine

INTERVENTIONS:
Procedure: Bilevel erector spinae plane block — Bilevel erector spinae plane block at 3rd and 5th thoracic vertebral levels
  Arms: Bilevel erector spinae plane block
Procedure: Single level erector spinae plane block — Single level erector spinae plane block at 5th thoracic vertebrae
  Arms: Single level erector spinae plane block
Drug: Intravenous morphine — Intravenous morphine 0.1 mg/kg
  Arms: Intravenous morphine

SUMMARY:
This study aims at comparing the analgesic efficacy and safety of bilevel erector spinae versus single level versus general anesthesia for breast cancer surgeries

ELIGIBILITY:
Inclusion Criteria:

* Female
* Diagnosed with breast cancer

Exclusion Criteria:

* Patient refusal
* coagulation defects
* bone metastases
* abnormal kidney and/or liver function tests

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Females
Enrollment: 126 (Actual)
Dates: Start 2022-06-27 (Actual); Primary Completion 2023-12-27 (Actual); Study Completion 2024-01-10 (Actual)

PRIMARY OUTCOMES:
Total analgesic requisite | First 24 hours postoperatively
  total postoperative morphine consumption

CONTACTS AND LOCATIONS:
Overall Officials: Walaa Y Elsabeeny, MD, Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- Walaa Y Elsabeeny, Cairo, Egypt